CLINICAL TRIAL: NCT06877897
Title: A Study of the Differences Between Submental Ultrasonography (SUS) and Assessment by Speech-Language Pathologists (SLP) for Nasogastric Tube Removal
Brief Title: Comparing the Assessment Accuracy Between Submental Ultrasound and Speech Therapists in Nasogastric Tube Removal
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 202411050RINC
Record Dates: First submitted 2025-03-04; First posted 2025-03-14 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Dysphagia Rehabilitation
Keywords: Nasogastric tube removal; Submental ultrasound; Acute dysphagia; Speech-language pathologist; hyoid bone displacement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SUS group (Experimental): The SUS group follows an oral feeding diet and tube removal training protocol based on submental ultrasound criteria, with a maximum hyoid bone displacement of ≥ 1.38 cm as an indicator of swallowing function.
  Interventions: Diagnostic Test: Submental ultrasound criteria
- SLP group (Active Comparator): The SLP group follows an oral feeding diet and tube removal training protocol based on the speech-language pathologist's assessment of swallowing function, which includes evaluating sensory and motor functions of the oral and facial muscles, phonation, swallowing motion, and other relevant factors.
  Interventions: Diagnostic Test: Routine swallowing function assessment of speech-language pathologist

INTERVENTIONS:
Diagnostic Test: Submental ultrasound criteria — According to the submental ultrasound criteria, a maximum hyoid bone displacement of ≥1.38 cm is required in the swallowing function assessment to qualify for the oral feeding diet and tube removal training protocol.
  Arms: SUS group
Diagnostic Test: Routine swallowing function assessment of speech-language pathologist — The speech-language pathologist (SLP) assessment includes the evaluation of sensory and motor functions of the oral and facial muscles, phonation, swallowing motion, and other relevant factors.
  Arms: SLP group

SUMMARY:
This randomized controlled trial aims to compare the assessment accuracy between submental ultrasound (SUS) and speech-language pathologists (SLP) for nasogastric tube removal in post-acute dysphagia adult patients. The primary question is whether the assessment accuracy of submental ultrasound (SUS) is equivalent to or better than that of speech-language pathologists (SLP).

Participants will undergo both submental ultrasound (SUS) and speech-language pathologists (SLP) assessments and will be randomly assigned to either the SUS group or the SLP group for further evaluation.

The SUS group will follow an oral feeding and tube removal training protocol based on submental ultrasound criteria for swallowing function (maximum hyoid bone displacement ≥ 1.38 cm). The SLP group will follow similar training protocols based on the speech-language pathologist's clinical assessment.

Researchers will compare outcomes such as nasogastric tube removal rate, vital signs, basic laboratory data, hyoid bone displacement on ultrasound, choking and aspiration rates, success rates of training protocols, and Functional Oral Intake Scale (FOIS) scores to determine if SUS is a reliable assessment method for swallowing function and NG tube removal.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and above
* Patients using a nasogastric tube
* Patients with a nasogastric tube placed due to acute conditions, such as increased oxygen demand, temporary loss of consciousness, or other illnesses causing weakness and a risk of aspiration. After treatment, there is no longer any indication for continued nasogastric tube placement.

Exclusion Criteria:

* Patients with impaired consciousness
* Patients with long-term nasogastric tube placement
* Patients requiring a high-concentration oxygen mask or mechanical ventilation with intubation
* Patients with significant drooling or frequent aspiration of saliva
* Patients who have undergone oral or head and neck surgery
* Patients who have received radiation therapy for the head and neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Comparing the assessment accuracy between submental ultrasound and speech therapist on nasogastric tube removal | From enrollment to the end of treatment at 8 weeks
  Rate of nasogastric tube removal Rate of successful completion of the tube removal training protocol

SECONDARY OUTCOMES:
Comparing the differences in ultrasound images between the submental ultrasound group and the speech therapist group | From enrollment to the end of treatment at 8 weeks
  Hyoid bone displacement (cm) during swallowing in submental images
Comparing the rate of aspiration pneumonia between the submental ultrasound group and the speech therapist group | From enrollment to the end of treatment at 8 weeks
  * of patients with chocking
  * of patients with aspiration pneumonia Vital signs: temperature in ℃, pulse in times/minute, respiratory rate: breaths per minute, blood pressure in mmHg, oxygen saturation in %

OTHER OUTCOMES:
Comparing the background information between the submental ultrasound group and the speech therapist group | From enrollment to the end of treatment at 8 weeks
  BMI in kg/m^2 Age in year Gender: male or female Indication for nasogastric tube usage
Comparing the GCS score between the submental ultrasound group and the speech therapist group | From enrollment to the end of treatment at 8 weeks
  Glasgow Coma Scale, score on the scale (3-15)
Comparing the Barthel index between the submental ultrasound group and the speech therapist group | From enrollment to the end of treatment at 8 weeks
  Barthel Index, score on the scale, 0 -100

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chung Shu, Doctor of Clinical Medicine, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hsu CY, Lai JN, Kung WM, Hung CH, Yip HT, Chang YC, Wei CY. Nationwide Prevalence and Outcomes of Long-Term Nasogastric Tube Placement in Adults. Nutrients. 2022 Apr 22;14(9):1748. doi: 10.3390/nu14091748. PMID 35565713
- [Result] Lee YS, Lee KE, Kang Y, Yi TI, Kim JS. Usefulness of Submental Ultrasonographic Evaluation for Dysphagia Patients. Ann Rehabil Med. 2016 Apr;40(2):197-205. doi: 10.5535/arm.2016.40.2.197. Epub 2016 Apr 25. PMID 27152268
- [Result] Allen JE, Clunie GM, Winiker K. Ultrasound: an emerging modality for the dysphagia assessment toolkit? Curr Opin Otolaryngol Head Neck Surg. 2021 Jun 1;29(3):213-218. doi: 10.1097/MOO.0000000000000708. PMID 33741822
- [Result] Hsiao MY, Chang YC, Chen WS, Chang HY, Wang TG. Application of ultrasonography in assessing oropharyngeal dysphagia in stroke patients. Ultrasound Med Biol. 2012 Sep;38(9):1522-8. doi: 10.1016/j.ultrasmedbio.2012.04.017. Epub 2012 Jun 12. PMID 22698507

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT06877897/Prot_SAP_001.pdf